CLINICAL TRIAL: NCT00574093
Title: 12 Months Case Series Open Study to Assess the Safety and Efficacy of Intravitreal Injection of Lucentis (Ranibizumab 0.5 mg)Used in Combination With Visudyne (Verteporfin PDT) in Naive Subjects With Subfoveal CNV Secondary to AMD
Brief Title: Efficacy and Safety Study of Lucentis (Ranibizumab) and Visudyne (Verteporfin) Combination Therapy in Neovascular AMD
Acronym: Luvi
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Monica Varano, Fondazione G.B. Bietti, IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBPD952AIT03
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Neovascular Age Related Macular Degeneration
Keywords: combination therapy; Lucentis; Visudyne
MeSH Terms: interventions — Ranibizumab; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): A: This will be a single arm study. Patients will be administered Lucentis™ on Day 1,at Months 1 and 2, and then as needed at intervals of at least 30 days through Month 11 based on the retreatment criteria algorithm. These patients will also be administered Visudyne® only on Day 3.
  Interventions: Drug: Ranibizumab; Verteporfin

INTERVENTIONS:
Drug: Ranibizumab; Verteporfin — Patients will be administered Lucentis™ 0.5 mg on Day 1, at Months 1 and 2, and then as needed at intervals of at least 30 days through Month 11 based on the retreatment criteria algorithm. These patients will also be administered Visudyne® only on Day 3.

SUMMARY:
This study is designed to evaluate the effect of Visudyne® combination therapy (Visudyne® [verteporfin for injection] and Lucentis™) on visual acuity outcomes. Study results will be submitted for publication to provide data that may help physicians refine the clinical management of patients with CNV secondary to age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This will be a single arm study. Patients will be administered Lucentis™ on Day 1, at Months 1 and 2, and then as needed at intervals of at least 30 days through Month 11 based on the retreatment criteria algorithm. These patients will also be administered Visudyne® only on Day 3.

Consenting patients will participate in the Screening Period to evaluate study eligibility. Patient eligibility assessments will include BCVA, contrast sensibility, speed reading and VFQ-25, a standard ophthalmic examination, OCT, color fundus photography, Fluorescein Angiography (FA), Green Indocyanine Angiography, Microperimetry and multifocal ERG.

BCVA and mean central retinal thickness measured by OCT will be repeated at every follow up visit.

Fluorescein Angiography (FA), Green Indocyanine Angiography, contrast sensibility and speed reading mean retinal sensitivity measured by microperimetry will repeated at month 3, 6, 9 and 12 month.

Color fundus photography at month 1, 3, 6, 9 and 12 month. Multifocal ERG will repeated at month 3 and 12 month. VFQ-25 will repeated at month 3 and 12.

The patient will receive ranibizumab monthly unless the BCVA got worse than 5 letters from the baseline BCVA and / or mean central retinal thickness evaluated with OCT increased less than 100 µm compared to month 2 visit (last date treatment). The repetition of the dose of ranibizumab should not begin before the thirtieth day following the end of the previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older male or female patients of any race with subfoveal CNV secondary to AMD (all types of lesion).
* The total area of CNV encompassed within the lesion must be >50% of the total lesion area. The total lesion area must have the greatest linear dimension ≤5400 microns (9 MPS Disc Areas).
* BCVA letter score in the study eye should be between 73 and 24 (approximately 20/40 to 20/320 Snellen Equivalent) using an ETDRS chart measured at 4 meters distance.

Exclusion Criteria:

* Any prior treatments with Visudyne, Macugen, Lucentis (Ranibizumab), Avastin (Bevacizumab) or other anti-angiogenic or corticosteroid intravitreal treatment in the study eye
* Prior external-beam radiation, subfoveal focal laser photocoagulation, transpupillary thermotherapy, pars plana vitrectomy in the study eye
* History of intraocular surgery in the study eye except for uncomplicated cataract surgery more than 90 days prior to treatment
* History of YAG-laser posterior capsulotomy in the study eye within 30 days prior treatment
* Use of non steroid antinflammatory drugs during the study
* Presence of angioid streaks, presumed ocular histoplasmosis syndrome, pathologic myopia (>8 D)
* Presence of fibrosis, haemorrhage, pigment epithelial detachments or other hypofluorescent lesions obscuring greater than 50% of the CNV lesion
* Tear (rip) of the retinal pigment epithelium
* Vitreal haemorrhage, retinal detachment or macular hole
* Epiretinal membrane
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with two or more topical pharmacological antiglaucomatous medication)
* Active or history of ocular inflammation or infection
* Aphakia and posterior capsule tear
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless they meet the following definition of postmenopausal
* Any systemic medical condition that may interferes with the safety of the patient
* Positive anamnesis for tumor in last the 5 years

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
the mean change from baseline in BCVA letters with ETDRS at Month 3,6,12. -the number of retreatments, the treatment-free interval and the % of retreated patients at month 3, 6, 12. -the mean retinal thickness change from baseline at month 3, 6 and 12. | 12 months

SECONDARY OUTCOMES:
% of patients that gain ≥5, ≥10, ≥15 letters BCVA; % of patients that lose <15 letters; Mean BCVA change and mean change of the total area of the lesion from baseline; Change of FA leakage; Mean retinal sensitivity change at month 3, 6 and 12 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Monica Varano, MD, Principal Investigator — Fondazione G.B. Bietti, IRCCS
Locations (1):
- Fondazione G.B.Bietti-IRCCS, Rome, Italy